CLINICAL TRIAL: NCT04054037
Title: A Study of APASL ACLF Research Consortium (AARC) Standards on Diagnosis and Treatment of Patients With Hepatic B Virus Related Acute on Chronic Liver Failure (HBV-ACLF) in China (AARC China Study)： a Multicentre Prospective Cohort Study
Brief Title: A Study of AARC Standards on Diagnosis and Treatment of Patients With HBV-ACLF in China (AARC China Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: AARC China Study
Record Dates: First submitted 2019-04-13; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Acute on Chronic Liver Failure; HBV
Keywords: APASL ACLF Research Consortium; Diagnosis and treatment standard; HBV-ACLF; acute on chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be restored in central lab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBV-ACLF Group: Patients with HBV related acute on chronic liver failure
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observation study, no intervention will be indicated during diagnosis and treatment.

SUMMARY:
The AARC China Study is to establish a widely recognized and harmonized standard of patients with HBV-ACLF in the Asia Pacific region.

DETAILED DESCRIPTION:
Acute on chronic liver failure (ACLF) is a clinically critical illness and has been extensively researched around the world. However, there is a potential "communication barrier" in the ACLF study; that is, different countries and regions, or different research collaboration groups, follow different ACLF definitions and related standards, making researchers in this field confuse in understanding the research value of relevant research and interpreting the research results. Important differences exist in the Asia-Pacific region and North America and Europe, such as the etiology, the clinical characteristics of the patient group, the requirements for cirrhosis, and the predisposing factors of the disease, making it necessary for China or the Asia-Pacific region to develop appropriate ACLF diagnosis standards and prognosis. In recent years, Chinese experts have also focused on the research progress of APASL ACLF Research Consortium (AARC) in the Asia-Pacific region. It is found that the AARC standards are more suitable for the diagnosis and treatment of patients with ACLF in China than the Western standards. The ACLF prediction model (TPPM model) established by Professor Qin.N's team predicts that the prognostic efficacy of patients with HBV-ACLF is significantly better than that of Western prognosis. The AARC China Study is to establish a widely recognized and harmonized standard of patients with HBV-ACLF in the Asia Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease: Chronic hepatitis B
* Acute deterioration of liver function: more than one of the below criteria

  1. development of new ascites within 4 weeks or re-emergence of ascites who have previous well controlled ascites (greater than or equal to grade 2 or 3; International ascites club criteria)
  2. development of hepatic encephalopathy
  3. development of gastrointestinal hemorrhage
  4. development of jaundice (serum bilirubin greater than or equal to 3mg/dl)
  5. development of bacterial infection
* spontaneous bacteremia: positive blood cultures without a source of infection
* spontaneous bacterial peritonitis: ascitic fluid polymorphonuclear cells >250/µL
* lower respiratory tract infections: new pulmonary infiltrate in the presence of: i) at least one respiratory symptom (cough, sputum production, dyspnea, pleuritic pain) with ii) at least one finding on auscultation (rales or crepitation) or one sign of infection (core body temperature >38_C or less than 36_C, shivering, or leukocyte count >10,000/mm3 or <4,000/mm3) in the absence of antibiotics
* Clostridium difficile Infection: diarrhea with a positive C. difficile assay
* bacterial entero-colitis: diarrhea or dysentery with a positive stool culture for Salmonella, Shigella, Yersinia, Campylobacter, or pathogenic E. coli;
* soft-tissue/skin Infection: fever with cellulitis
* urinary tract infection (UTI): urine white blood cell >15/high-power field with either positive urine gram stain or culture;
* intra-abdominal infections: diverticulitis, appendicitis, cholangitis, etc.
* other infections not covered above;
* fungal infections as a separate category.

Exclusion Criteria:

* Patients who do not have chronic liver disease
* Patients who have hepatocellular carcinoma
* Patients who admitted for extrahepatic manifestations
* Patients who have HIV infection
* Patients who admitted for symptomatic control of chronic liver disease, other than acute deterioration of liver function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HBV-related acute-on-chronic liver failure
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Non-liver transplant mortality | 30 days, 90 days
  Non-liver transplant mortality rate at 30 days, 90 days

SECONDARY OUTCOMES:
progression of Chronic liver disease | 3 years
  Incidence of liver disease progression (such as cirrhosis, decompensation of liver function, liver cancer, liver transplantation, or liver related death)

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, MD., PhD., Study Director — Department of Infectious Disease, Tongji Hospital
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided